CLINICAL TRIAL: NCT05862636
Title: Who Fares Best With Mindfulness Meditation - Understanding the Individual Effects of Mindfulness
Brief Title: Who Fares Best With Mindfulness Meditation
Status: Recruiting | Type: Observational
Sponsor: Prof. dr. Filip Raes (Other)
Collaborators: University of Exeter (Other)
Responsible Party: Sponsor-Investigator, Prof. dr. Filip Raes, Professor, KU Leuven
Organization: KU Leuven (Other)
Other Study IDs: s66664; IRAS ID 313533 (Other: Health Research Authority UK)
Record Dates: First submitted 2023-01-31; First posted 2023-05-17 (Actual); Last update posted 2025-01-06 (Actual); Status verified 2025-01

CONDITIONS: Healthy; Depression; Mental Health Issue
MeSH Terms: conditions — Depression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Mindfulness centre for general public: Mindfulness course attenders at a mindfulness centre that offers mindfulness trainings for the general public. Participants are thus not selected based on any complaints they may have.
  Interventions: Behavioral: Mindfulness Training
- Stress clinic: Mindfulness course attenders at a stress clinic associated with a hospital that offers mindfulness courses for participants with mild complaints, such as stress or worry.
  Interventions: Behavioral: Mindfulness Training

INTERVENTIONS:
Behavioral: Mindfulness Training — All participants will follow a mindfulness course consisting of group sessions of 2-3h duration that are organized (nearly) weekly and are spread over a period of eight weeks. The specific timeline and organisation of the course may differ between the participating sites but all courses will involve a comparable amount of contact hours with the mindfulness trainer. Each session consists of guided experiential mindfulness exercises (e.g., body scan, breathing space, breath focus, walk meditation), sharing of experiences of these exercises, reflections in small groups, psychoeducation, and review of home practices.
  The mindfulness courses are based on one of the two most well-known MBIs, Mindfulness-Based Cognitive Therapy (Segal et al., 2002) and Mindfulness-Based Stress Reduction (Kabat-Zinn, 1990), or a combination thereof. Courses follow a standardised protocol with group sessions and daily homework tasks taught by experienced and certified mindfulness trainers.

SUMMARY:
The overall aim of this observational study is to investigate how individual differences influence the effects of mindfulness meditation to uncover for whom mindfulness is beneficial and for whom it may be harmful. The first objective is to identify the mechanisms underlying the effects of mindfulness meditation on mental health. The second objective is to examine how three candidate factors, namely trauma symptoms, tendency to dissociate, and repetitive negative thinking, influence the effect of mindfulness meditation on mental health.

Adults who enrolled for a Mindfulness-Based Intervention (MBI) at the participating sites (n=120 in total) will be invited to participate. Before the start of the MBI, after half of the sessions, at the end of the MBI and at 3-months follow-up, participants will complete self-report questionnaires. The main outcomes are symptoms of anxiety and depression, quality of life, wellbeing, and adverse effects resulting from the MBI. A subset of participants will be invited for a semi-structured interview after the end of the intervention.

Update December 2024:

Instead of analysing all subsamples recruited from the different sites separately, the investigators will now analyse all participants from all sites jointly. This amendment has two reasons. First, analysing all participants jointly allows to statistically compare the differences in effects across sites by including a variable that indicates from which site a participant was recruited. If the subsamples are analysed separately, the investigators can only compare the results at face-value but cannot determine whether the effects are statistically different across sites. Second, recruitment could not start at one site because of a restructuring of the mindfulness interventions there and the investigators are experiencing recruitment difficulties in a second site (recruited 5 participants within 1.5 years). Thus, it will not be feasible to recruit 120 participants per site. For those two reasons, the investigators decided to analyse all participants jointly and only recruit 120 participants in total for the quantitative part of this study (see updated study protocol).

DETAILED DESCRIPTION:
This project aims to investigate how individual differences influence the effects of mindfulness meditation to gain a first understanding of the personalised effects of mindfulness and uncover for whom mindfulness is beneficial and for whom it may be harmful. In a first step towards a better understanding of the effects of mindfulness mediation on each individual, the investigators aim to identify the mechanisms underlying the effects of mindfulness meditation on mental health and wellbeing (first objective). Based on prior research, the investigators hypothesise that mindfulness meditation exerts its effects via internal awareness, decentering, and non-judgment, but the investigators will also explore other mindfulness skills as potential mechanisms. Knowing the underlying mechanisms will help understand why mindfulness meditation leads to improved mental health in some individuals while it may lead to harm in other individuals. In a second step, the investigators aim to examine specific characteristics of individuals that may influence whether mindfulness meditation has beneficial or possibly harmful effects. Specifically, the investigators aim to examine how three candidate factors, namely trauma symptoms, tendency to dissociate, and repetitive negative thinking, influence the effect of mindfulness meditation on mental health and wellbeing (second objective). Knowing how these individual characteristics influence the effect of mindfulness meditation will clarify for whom mindfulness works best and for whom it may lead to undesired effects.

For both objectives, mental health and wellbeing will be measured using self-report questionnaires to determine the effects of the mindfulness intervention on participants' mental health and wellbeing. To achieve the first objective, the investigators will measure change of different mindfulness skills (the hypothesised mechanisms) with self-report questionnaires across the mindfulness intervention in order to test whether the mindfulness intervention leads to change in mindfulness skills, which in turn leads to change in outcomes. To achieve the second objective, the investigators will measure baseline levels of candidate factors with self-report questionnaires in order to test whether these candidate factors influence in what way the mindfulness intervention affects mental health and wellbeing. Candidate factors are trauma history and symptoms, tendency to dissociate, and repetitive negative thinking. Additionally, the investigators will measure obsessive-compulsive disorder related beliefs as potential candidate factors, as these beliefs influenced the effects of mindfulness in our own clinical practice. Meditation practice-related variables such as frequency, intentions and previous experience will be measured in order to control for potential practice-related effects on mental health.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in a mindfulness-based intervention at one of the participating sites

Exclusion Criteria:

* Insufficient knowledge of the Dutch or English language (depending on the study site)
* No internet access

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults who enrolled for a Mindfulness-Based Intervention (MBI) at one of the participating study sites.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2023-02-21 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Change in Patient Health Questionnaire-4 (PHQ-4) | Before the MBI, 4-weeks after start of MBI, 8 weeks after start of MBI, and 3 months after the end of the MBI
  The PHQ-4 is a 4-item scale that measures symptoms of depression and anxiety over the last two weeks. Items are scored on a 4-point Likert scale ranging from 0 (not at all) to 3 (nearly every day).
Change in Recovering Quality of Life (ReQol-10) | Before the MBI, 4-weeks after start of MBI, 8 weeks after start of MBI, and 3 months after the end of the MBI
  The ReQol-10 is a 10-item scale that measures quality of life over the last week. Items are scored on a 5-point Likert scale ranging from 0 (none of the time) to 4 (most or all of the time).
Change in Short Warwick-Edinburgh Mental Well-being Scale (SWEMWBS) | Before the MBI, 4-weeks after start of MBI, 8 weeks after start of MBI, and 3 months after the end of the MBI
  The SWEMWBS is a 7-item scale that measures wellbeing over the last two weeks. Items are scored on a 5-point Likert scale ranging from 1 (none of the time) to 5 (all of the time).
Change in Meditation-Related Adverse Effects Scale, Mindfulness-Based Program version (MRAES-MBP) | Before the MBI, 4-weeks after start of MBI, 8 weeks after start of MBI, and 3 months after the end of the MBI
  The MRAES-MBP is a 14-item scale that measures mindfulness-related adverse events over the last four weeks. Items are scored on a 5-point Likert scale ranging from 1 (never) to 5 (very often).

SECONDARY OUTCOMES:
Subjective experience of mindfulness practice effects assessed during interview | 8 weeks after start of MBI
  Subjective experience of the impact of mindfulness practice on participants' lives and what factors contributed to their experience of mindfulness practice.
Change in Comprehensive Inventory of Mindfulness Experiences - Short Form (CHIME-SF) | Before the MBI, 4-weeks after start of MBI, 8 weeks after start of MBI, and 3 months after the end of the MBI
  The CHIME-SF is a 24-item scale that measures mindfulness skills over the last two weeks. Items are scored on a 6-point Likert scale ranging from 1 (never or almost never) to 6 (always or almost always).
Brief Dissociative Experiences Scale (DES-B) | Before the MBI
  The DES-B is a 8-item scale that measures participants' tendency to dissociate. Items are scored on a VAS scale ranging from 0% (never) to 100% (always).
Perseverative Thinking Questionnaire (PTQ) | Before the MBI
  The PTQ is a 15-item scale that measures repetitive negative thinking. Items are scored on a 5-point Likert scale ranging from 0 (never) to 4 (almost always).
Modified version of the Life Events Checklist for DSM-5 (LEC-5) | Before the MBI
  The LEC-5 is a 17-item scale that measures exposure to traumatic events. Items are scored as either yes (happened to you, you witnessed it, you learned about it happening to a close friend or family member, or you were exposed to it as part of your job) or no (event does not apply to you).
International Trauma Questionnaire (ITQ) | Before the MBI
  The ITQ is a 18-item scale that measures PTSD symptoms. Items are scored on a 5-point Likert scale ranging from 0 (not at all) to 4 (extremely).
Obsessive Beliefs Questionnaire (OBQ-9) | Before the MBI
  The OBQ-9 is a 9-item scale that measures obsessive-compulsive disorder related beliefs. Items are scored on a 7-point Likert scale ranging from 1 (disagree very much) to 7 (agree very much).

OTHER OUTCOMES:
Previous experience with meditation | Before the MBI
  An 8-item scale measuring participants' previous experience with meditation including duration of practice and frequency of practice during the last 4 weeks.
Frequency of mindfulness home practice | 4-weeks after start of MBI, 8 weeks after start of MBI, and 3 months after the end of the MBI
  A 4-item scale measuring frequency and duration of home practice during the last 4 weeks.
Change in Practice Quality-Mindfulness (PQ-M) | 4-weeks after start of MBI, 8 weeks after start of MBI, and 3 months after the end of the MBI
  The PQ-M is a 6-item scale that measures quality of mindfulness practice during the last meditation session. Items are scored on a VAS scale ranging from 0% (the statement reflects my experience none of the time) to 100% (the statement reflects my experience all of the time).
Intentions of meditation practice | 4-weeks after start of MBI, 8 weeks after start of MBI, and 3 months after the end of the MBI
  A 2-item scale measuring intentions for meditation practice on a 7-point Likert scale ranging from "never" to "every time I meditate".
Modified version of the Credibility/ Expectancy Questionnaire (CEQ) | Before the MBI, 4-weeks after start of MBI, 8 weeks after start of MBI, and 3 months after the end of the MBI
  The CEQ is a 4-item scale that measures training expectancy. Items are scored on a 9-point Likert scale ranging from 1 (not at all) to 9 (very much).
Session attendance | 8 weeks after start of MBI
  A 2-item scale measuring number of attended sessions and drop-out.

CONTACTS AND LOCATIONS:
Overall Officials: Filip Raes, Prof. dr., Principal Investigator — KU Leuven
Locations (3):
- Belgium (2):
  - ZNA Stresskliniek, Antwerp
  - Mindful Me, Deinze
- AccEPT clinic, Exeter, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Moderately sensitive information including age, demographic data, all other data coming from questionnaires and interview transcripts will be pseudonymized and shared with other researchers upon request. This dataset will only comprise data of those participants who agreed to their data being shared on the consent form.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: The coded, pseudonymized dataset and supporting information (see above) will be available beginning from 3 months and ending 10 years after publication of the research results.
Access Criteria: The receiving party will be bound by contractual agreement to keep the transferred data confidential at all times, to only process the data for the purpose of the Study or for improving scientific knowledge about mindfulness and is not permitted to link the data with other data which might render the information more identifiable. To this end, appropriate Data Transfer Agreements (DTAs) will be established.

DOCUMENTS (2):
  • Study Protocol (2024-12-06): https://cdn.clinicaltrials.gov/large-docs/36/NCT05862636/Prot_001.pdf
  • Statistical Analysis Plan (2024-12-23): https://cdn.clinicaltrials.gov/large-docs/36/NCT05862636/SAP_002.pdf